CLINICAL TRIAL: NCT02887703
Title: Augmenting Balance in Individuals With Cerebellar Ataxias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kathleen Sienko (Other)
Responsible Party: Sponsor-Investigator, Kathleen Sienko, Associate Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00116756
Record Dates: First submitted 2016-08-22; First posted 2016-09-02 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Cerebellar Ataxia
Keywords: ataxia; balance training; vibrotactile biofeedback; sensory augmentation; cerebellar ataxia
MeSH Terms: conditions — Cerebellar Ataxia; Ataxia | interventions — Haptic Technology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensory Augmentation Group 1 (Experimental): Each subject in Group 1 will undergo 6 weeks of balance training with sensory augmentation followed by 6 weeks of balance training without sensory augmentation.
  Interventions: Behavioral: Sensory Augmentation
- Sensory Augmentation Group 2 (Experimental): Each subject in Group 2 will undergo 6 weeks of balance training without sensory augmentation followed by 6 weeks of balance training with sensory augmentation.
  Interventions: Behavioral: Sensory Augmentation

INTERVENTIONS:
Behavioral: Sensory Augmentation — Sensory augmentation is a technique of augmenting or replacing compromised sensory information. In the context of sensory-based balance impairments, a sensory augmentation device provides cues of body motion that supplement an individual's remaining intact sensory systems.
  Other Names: vibrotactile biofeedback; haptic feedback

SUMMARY:
This study evaluates the effectiveness of a 12-week in home balance training program with and without sensory augmentation for individuals with ataxia. Subjects wear a belt while performing balance exercises three times per week for 12 weeks. The belt measures body motion and has small vibrating elements called tactors mounted inside that when turned on, feel like a cell phone set to vibrate. The tactors provide information about body motion and indicate when and how to make a postural correction. Subjects will receive six weeks of balance training with the tactors turned on and six weeks of balance training with the tactors turned off.

DETAILED DESCRIPTION:
Cerebellar ataxias are a group of degenerative neurological disorders, resulting in deficits in speech, limb control, balance, and gait. Individuals with degenerative cerebellar ataxias are at a high-risk of falling and have progressive impairments in motor coordination resulting in unsteadiness in gait and posture. No definitive treatment options are available for ataxia. There is therefore a critical need to identify strategies to improve motor function and reduce falls in patients with ataxia. Physical therapy has been demonstrated to improve motor function in subjects with cerebellar ataxia, but the gains in performance following balance training are modest. Sensory augmentation is a technique of augmenting or replacing compromised sensory information. In the context of sensory-based balance impairments, a sensory augmentation device provides cues of body motion that supplement an individual's remaining intact sensory systems. The investigators hypothesize that sensory augmentation may improve the effectiveness of balance training in individuals with ataxia, and aid in greater improvement in motor function than traditional physical therapy alone. Sensory augmentation has been shown to decrease body sway during real-time operation in a laboratory setting in individuals with vestibular deficits and peripheral neuropathy, and general age-related declines in balance performance. Preliminary results suggest that persistent improvements in balance performance exist over time periods of hours to days following a small number of training sessions. This study aims to characterize the effects of sensory augmentation in individuals with ataxia during static and dynamic balance exercises over a period of twelve weeks of in home balance training with and without vibrotactile sensory augmentation.

ELIGIBILITY:
Inclusion Criteria:

* Report to be in good general health
* Are able to read and comprehend English
* Have been diagnosed with either an inherited or sporadic degenerative cerebellar or sensory ataxia
* Are able to stand for at least 30 seconds with no support
* Must be willing and able to comply with study schedule
* Must have wireless internet (WiFi) enabled in their home
* Must be able to perform the home based exercises safely (as assessed by clinical research staff)

Exclusion Criteria:

* Are pregnant or believe subject might be pregnant
* Have been diagnosed with arthritis or other musculoskeletal disorder affecting joints, muscles, ligaments and/or nerves that affects the way subject moves
* Have a history of fainting
* Have a severe vision or hearing impairment that is not corrected by glasses or hearing aids
* Have sustained a fall in the last six months that resulted in hospitalization or serious injury
* Have corrected vision worse than 20/70 (considered threshold for moderate visual impairment)
* Are unable to feel the vibrotactile feedback on their torso through the standard t-shirt provided by the study team
* Have ankle dorsi-flexor/plantar-flexor weakness as demonstrated < 4/5 on manual muscle test
* Have limited ankle range of motion demonstrated by inability to dorsiflex to neutral with the knee extended
* Report lower extremity fracture/sprain in the past six months or more than one lower extremity total joint replacement
* Are medically unstable (e.g. chest pain upon exertion, dyspnea, infection)
* Have a history of any other neurological disease besides ataxia that might affect balance (e.g. cerebral vascular accident, Parkinson's disease, MS, ataxia)
* Have a body mass index (BMI) over 30 kg/m2, computed from subject height and weight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Scale for the assessment and rating of ataxia (SARA) | pre balance training (week 1), mid balance training (week 6), post balance training (week 12)
  An 8-item scale including walking, standing, sitting, nose-to-finger movements, and fast alternating movements. Standard assessment scale for determining impairment level in individuals with ataxia.

SECONDARY OUTCOMES:
Change in 10-meter Preferred Gait Speed | pre balance training (week 1), mid balance training (week 6), post balance training (week 12)
  Preferred gait velocity will be measured while walking a 10-meter path.
Change in 10-meter Fast Gait Speed | pre balance training (week 1), mid balance training (week 6), post balance training (week 12)
  Fast gait velocity will be measured while walking a 10-meter path.

OTHER OUTCOMES:
Change in Five Times Sit to Stand Test | pre balance training (week 1), mid balance training (week 6), post balance training (week 12)
  A stop watch is used to measure how long it takes a participant to stand up and sit down five times in a row without using their hands.
Change in Activities Specific Balance scale (ABC) | pre balance training (week 1), mid balance training (week 6), post balance training (week 12)
  A 16-item questionnaire for participants to self report their balance confidence during activities of daily living.
Change in Berg Balance Score | pre balance training (week 1), mid balance training (week 6), post balance training (week 12)
  A 14-item scale to assess balance including sit-to-stand, standing, turning and picking up items from the floor.
Change in Dynamic Gait Index (DGI) | pre balance training (week 1), mid balance training (week 6), post balance training (week 12)
  An 8-item test to evaluate gait function including normal and fast walking, changing speeds, stepping over obstacles, pivoting, walking with head turns, and stairs.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen H Sienko, Ph.D., Principal Investigator — Department of Mechanical Engineering
Locations (1):
- Department of Mechanical Engineering, University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided